CLINICAL TRIAL: NCT07098429
Title: A Comparison Of Postoperative Pain With And Without Instillation Of Bupivacaine During Laparoscopic Cholecystectomy
Brief Title: Postoperative Pain After Instillation Of Bupivacaine During Laparoscopic Cholecystectomy
Acronym: BUPA-LC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Recep Tayyip Erdogan Hospital Pakistan (Other)
Responsible Party: Principal Investigator, Noman Yousaf, Noman Yousaf, Indus Hospital and Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHHN _IRB_2024_04_002
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Laparoscopic Cholecystectomy; Post Operative Analgesia; Bupivacaine
Keywords: Laparoscopic Cholecystectomy Analgesia; Gallstones; Outcomes; Postoperative Pain
MeSH Terms: conditions — Gallstones; Pain, Postoperative | interventions — Postoperative Period; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline Group (Placebo Comparator): In 30 patients who underwent Laparoscopic Cholecystectomy , 20ml of 0.9% normal saline instillation in gallbladder fossa after removal of gallbladder
  Interventions: Drug: Bupivacain (Postoperative); Drug: Normal (0.9%) saline
- Bupivacaine Group (Experimental): In 30 patients who underwent Laparoscopic Cholecystectomy , 20ml of 0.25% Bupivacaine instillation in gallbladder fossa after removal of gallbladder
  Interventions: Drug: Bupivacain (Postoperative)

INTERVENTIONS:
Drug: Bupivacain (Postoperative) — 20ml of 0.25% bupivacaine instillation in gallbladder fossa after removal of gallbladder in laparoscopic cholecystectomy this study used less amount of drug
Drug: Normal (0.9%) saline — In 30 patients who underwent Laparoscopic Cholecystectomy , 20ml of 0.9% normal saline instillation in gallbladder fossa after removal of gallbladder.
  Arms: Normal Saline Group

SUMMARY:
This study aims to compare the level of postoperative pain experienced by patients undergoing laparoscopic cholecystectomy with and without the use of intraperitoneal bupivacaine. Bupivacaine, a long-acting local anesthetic, is hypothesized to reduce postoperative pain when instilled into the peritoneal cavity at the end of the procedure. The study will involve adult patients undergoing elective laparoscopic cholecystectomy and will assess pain levels using standardized pain scoring methods at various postoperative intervals. By evaluating and comparing outcomes in both groups, the study seeks to determine whether the routine use of intraperitoneal bupivacaine provides significant analgesic benefits, contributing to enhanced recovery and improved patient comfort following surgery

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is now widely regarded as the standard treatment for gallstones due to its advantages over open surgery, including reduced postoperative pain, shorter hospital stays, and quicker recovery. Despite these benefits, many patients still experience significant pain after surgery, attributed to factors such as port-site incisions and the residual gas used during the procedure. This study was designed to assess whether the use of bupivacaine, a local anesthetic instilled into the gallbladder bed during surgery, can help in reducing postoperative pain. The objective was to compare the pain levels in patients who received bupivacaine with those who received a placebo (normal saline) during LC.

The study included both male and female patients between the ages of 14 and 70 who were scheduled for elective laparoscopic cholecystectomy. Patients were excluded if they had a known allergy to bupivacaine, were pregnant or breastfeeding, had acute cholecystitis or gallbladder empyema, or if their surgery was converted from laparoscopic to an open procedure. A total of 60 patients were enrolled and randomly divided into two groups. Group A received 20 ml of 0.25% bupivacaine instilled into the gallbladder fossa after gallbladder removal, while Group B received 20 ml of normal saline. Both groups also received standard local anesthesia at the port sites. Following surgery, pain levels were recorded at 1, 3, 6, 12, and 24 hours using a standard pain scoring system. Additionally, the time to the first request for rescue analgesia was documented.

Participants in this study might benefit from reduced postoperative pain, decreased need for additional analgesics, and a potentially quicker recovery. The risks associated with participation were minimal, limited primarily to rare allergic reactions or local discomfort due to bupivacaine. Importantly, no narcotics were used, thereby reducing risks related to sedation or dependency.

The study was conducted at Recep Tayyip Erdogan Hospital in Muzaffargarh, Pakistan. It commenced on 19 November 2024 and concluded on 10 April 2025, with a total duration of approximately five months. The authors of the study declared that no external funding was received

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, having age 14-70 years, admitted to undergo scheduled Laparoscopic Cholecystectomy

Exclusion Criteria:

Patients with history of hypersensitivity to bupivacaine Acute cholecystitis Pregnancy Lactating mothers Empyema of the gallbladder and laparoscopic converted to open surgery

-

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Pain Assessment after Laparoscopic Cholecystectomy | Pain assessment at 1st 3rd 6th 12th and 24th hour
  After instillation of drug, pain assessment will be done using Wong Baker Faces

CONTACTS AND LOCATIONS:
Overall Officials: Noman Yousaf, MBBS, Principal Investigator — Indus Hospital & health Network
Locations (1):
- Recep Tayyip Erdogan Hospital, Muzaffargarh, Pakistan, Muzaffargarh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No